CLINICAL TRIAL: NCT06901739
Title: New Dietary Intervention Strategies on the Intestinal Microbiota to Improve Mental Health Subjects With Obesity: Therapeutic Potential of a Synbiotic.
Brief Title: Therapeutic Potential of a Synbiotic to Improve Mental Health in Subjects With Obesity.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Celia Bañuls (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Celia Bañuls, Principal Investigator, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Organization: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PI24/01010
Record Dates: First submitted 2025-03-23; First posted 2025-03-30 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Obese Patients (BMI ≥ 30 kg/m²); Anxiety; Depressive Disorder
Keywords: Microbiota; Inflammation; Symbiotic; Tannins; Mental disorders; Obesity
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder; Inflammation; Mental Disorders; Obesity | interventions — Synbiotics; Tannins; Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Synbiotic supplement in subjects with obesity and mental disorders (Experimental): Subjects with both obesity and mental disorders (only including anxiety or depression diagnosed disorders) will recieve the synbiotic supplement and nutritional intervention by a registered dietitian for 12 weeks.
  Interventions: Dietary Supplement: Synbiotic
- Synbiotic supplement in subjects with obesity and without mental disorders (Active Comparator): Subjects with obesity yet without diagnosed mental disorders will recieve the synbiotic supplement and nutritional intervention by a registered dietitian for 12 weeks.
  Interventions: Dietary Supplement: Synbiotic
- Placebo in subjects with obesity and mental disorders (Placebo Comparator): Subjects with both obesity and mental disorders will recieve nutritional intervention by a registered dietitian and a supplement containing a powder with an identical color compared to the synbiotic supplement.
  Interventions: Dietary Supplement: Placebo
- Placebo in subjects with obesity and without mental disorders (Placebo Comparator): Subjects with both obesity but no diagnosed mental disorders will recieve nutritional intervention by a registered dietitian and a supplement containing a powder with an identical color compared to the synbiotic supplement.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Synbiotic — The synbiotic supplement contains both tannins (350mg) and probiotic strains (Lactobacillus acidophilus, Lactobacillus casei, y Bifidobacterium lactis 2×10 9 UFC/g each) that have already demonstrated a positive health effect in obesity. Besides, participants will follow a dietary intervention to improve their dietary habits and reduce weight by a registered dietitian.
  Other Names: tannins; probiotic
  Arms: Synbiotic supplement in subjects with obesity and mental disorders; Synbiotic supplement in subjects with obesity and without mental disorders
Dietary Supplement: Placebo — Subjects will recieve a placebo supplement, contained in an identical capsule form as the synbiotic, along with the same dietary intervention to improve their dietary habits and reduce weight by a registered dietitian.
  Arms: Placebo in subjects with obesity and mental disorders; Placebo in subjects with obesity and without mental disorders

SUMMARY:
Obese individuals are a particularly vulnerable population for mental health problems, especially depression and anxiety. The aim of this study is to evaluate whether the intake of a synbiotic, composed of prebiotics and beneficial intestinal bacterial strains, is capable of producing changes in the gut microbiota and its functionality, improving metabolic and inflammatory parameters, intestinal function and appetite control in patients with obesity and psychological disorders. In addition, the production of neurotransmitters at the level of the gut-brain axis will be studied, as well as mood and quality of life. For this purpose, a prospective, randomized, doubleblind, placebo-controlled intervention study will be carried out in patients with obesity (BMI=30-40 kg/m2) and symptoms of anxiety and/or depression, or patients with obesity but without these psychological disorders (n=120). The groups will be randomly divided into two groups (n=60) according to the intake of a synbiotic (1 capsule/day composed of bifidobacterium, Lactobacillus and tannin-based phytocomplexes) or its corresponding placebo for 12 weeks. Individualized psychological and nutritional follow-up will be carried out, demographic, lifestyle and mental health variables will be collected, and biological samples will be collected before and after the intervention. In addition, all patients will undergo an assessment of body composition and nutritional status, together with cardiovascular risk factors and comorbidities (hypertension, dyslipidemia, DM2, insulin resistance). Inflammatory parameters (IL6, TNF , IL1b, adiponectin, PAI-1, IL10, resistin, adipsin), antioxidant capacity, intestinal function (zonulin, LPS, occludin, LBP, FABP2/I-FABP, -glucan, Reg3A), satiety, appetite control (Leptin, GLP1, GIP, Ghrelin, PP) and neurotransmitter production (cortisol, dopamine, serotonin, oxytocin) in plasma/serum, urine or saliva using ELISA Kits and Luminex XMAP technology will be analyzed. In addiition, the investigators will perform analysis of genetic markers of inflammatory and metabolic pathways (Nanostring technology), metabolomic profiling (NMR spectroscopy and PLS-DA) in plasma, and both content and diversity of the intestinal microbiota (16S rRNA amplicons, and direct metagenomic sequencing, with Illumina MiSeq technology) in faeces will be evaluated.

Finally, the investigators will study in vitro the mechanism of action of colonic digest on complex cellular models that simulate the gut-brain axis (organ-on-chip model, OoC).

DETAILED DESCRIPTION:
Obesity is one of the most widespread chronic diseases globally, resulting from a complex interaction between dietary habits and environmental and genetic factors. According to the statistics from the World Health Organization, more than 1.9 billion adults are overweight, and approximately 650 million people suffer from obesity. Moreover, these individuals are at a higher risk of developing numerous metabolic disorders, such as type 2 diabetes, atherosclerosis, cardiovascular diseases, non-alcoholic fatty liver disease, reproductive issues, and some forms of cancer. Lifestyle and pharmacological interventions are two of the most important strategies for treating obesity. However, strict lifestyle changes are often only accepted by a limited number of individuals, and anti-obesity drugs can have some adverse effects, while their efficacy is often diminished after prolonged use. Therefore, a significant unmet need is the lack of convenient and effective adjunctive therapies for treating obesity.

There is a bidirectional association between obesity and mood disorders such as depression and anxiety. Obesity also has a negative effect on health and quality of life, as well as on self-esteem. Specifically, it is estimated that approximately 50% of individuals with obesity develop depressive and anxious traits, which are more common in females and more frequent as the degree of obesity increases. Furthermore, people with obesity often suffer a considerable emotional burden, increasing stress, daily worries, and even experiencing difficulties in performing daily life activities. Added to the stigma of the disease, which has a negative impact on self-esteem and body image, this worsens the quality of life and emotional state of these individuals. Therefore, mental health is closely interconnected with obesity, and addressing both the physical and emotional aspects is crucial for promoting overall well-being. It is important to adopt a holistic approach that includes interventions in diet, physical exercise, and emotional and psychological support for those struggling to maintain a healthy weight and adequate mental health.

The gut-brain axis is a bidirectional communication network between the gut and the central nervous system, functioning through neuroimmune and neuroendocrine processes. Its involvement in the onset of depression has been postulated and is mediated by molecules such as short-chain fatty acids, gamma-aminobutyric acid (GABA), and tryptophan metabolites originating from the gut microbiota. In situations of dysbiosis or alterations in microbiota homeostasis, the gut-brain pathways can be found deregulated and are associated with neuroinflammation and altered blood-brain barrier permeability. Moreover, alterations in the gut microbiota may contribute to a depressive state by directly affecting the release of neurotransmitters such as serotonin and dopamine, influencing the stress response and the hypothalamic-pituitary-adrenal (HPA) axis, affecting brain-derived neurotrophic factor (BDNF) levels, and triggering the release of inflammatory cytokines. For example, depression is associated with an increased release of C-reactive protein (CRP) and cytokines such as IL-1, IL-2, IL-6, IFN-y, and IL-1ß.

Obesity also causes inflammation at the intestinal level, insulin resistance, and body fat deposits. Research in this field suggests that there is a bidirectional relationship between the composition of the gut microbiota, obesity, and insulin resistance. It has been observed that people with obesity have a different microbial composition compared to those with a healthy weight. It is believed that this alteration in the gut microbiota could further contribute to the progression of obesity by increasing the ability to extract energy from food, promoting low-grade inflammation, increasing lipogenesis, decreasing fatty acid oxidation, and increasing triglyceride accumulation at the hepatic level, among other mechanisms.

Considering the role of the gut microbiota in regulating the immune system and inflammation, it can be observed that chronic inflammation is linked to both obesity and psychological disorders, including depression and anxiety. These changes in the gut microbiota may contribute to systemic inflammation and immune dysfunction, which in turn could affect both obesity and psychological disorders. Some gut bacteria can produce neurotransmitters that are absorbable at the intestinal level, such as serotonin or GABA, which are important for regulating mood and anxiety. It is believed that changes in the composition of the gut microbiota could affect the production of these neurotransmitters, and therefore, influence mental health.

Although lifestyle modifications, such as caloric restriction and physical exercise, are considered the best therapies for weight loss, there are other adjunctive options, such as the modulation of the gut microbiota, that could be useful for people with obesity. Studies in which prebiotics, probiotics, and synbiotics were administered to individuals with obesity have shown their beneficial effects on weight reduction and other metabolic parameters through the modulation of the gut microbiota. Due to the emerging evidence implicating the gut-brain axis in obesity and its relation to psychological disorders, there has been increased interest in the development of these treatments as therapies for restoring the gut microbiota.

Prebiotics are functional foods, given their beneficial role in promoting health and preventing disease. An example is tannins, considered bioactive compounds due to their ability to modulate metabolic processes and promote health. Much of the tannins ingested reach the large intestine, where the gut microbiota converts them into metabolites, including short-chain fatty acids such as acetate, propionate, and butyrate. These short-chain fatty acids are important metabolites that can have various beneficial effects on the host's intestinal and overall health. They also exert a potential antidiabetic effect through the following mechanisms: (i) Improvement of insulin and proinsulin levels in the blood: the affinity of tannins for binding to polysaccharides causes a delay and a decrease in the availability of glucose in the gastrointestinal tract. Additionally, several studies have reported the potential for inhibiting the activities of α-amylase and α-glucosidase through hydrolyzable tannins and condensed tannins, respectively. (ii) Insulin-like effect on insulin-sensitive tissues: procyanidins may act on specific components of the intracellular insulin signaling pathway. (iii) Regulation of the antioxidant environment of pancreatic cells: oxidative stress is believed to play a role in insulin resistance as it determines pancreatic cell apoptosis. Additionally, the expression of genes related to antioxidant enzymes in the pancreas is low. The high antioxidant capacity of tannins can counteract the pathogenesis of insulin resistance, along with their anti-inflammatory properties (they decrease TNFα, IL-1, IL-6 levels, etc.) and cardioprotective properties (they increase superoxide dismutase, decrease ROS, etc.).

Specifically, high molecular weight tannins reach the gut microbiota in the colon showing a prebiotic effect. In this case, the compounds are metabolized by microorganisms, producing metabolites with different bioavailability, activity, or functional effects compared to the original molecule. Finally, tannins can modulate the composition and function of the gut microbiota, selectively inhibiting pathogens and promoting the growth of beneficial bacteria.

Probiotics are preparations of microorganisms that, when administered in appropriate conditions and amounts, improve the microbial balance of the gut. These microorganisms have been shown to suppress inflammation and modulate the immune system by preventing the induction of the IL-8 cytokine in the human colon epithelium, as well as reducing intestinal permeability, inhibiting endotoxemia. Probiotic interventions can contribute to the treatment of obesity and associated complications by improving the abundance and function of the gut microbiota. Therefore, the combination of prebiotic and probiotic interventions (synbiotics) can provide a synergistic and effective therapy for metabolic disorders. Additionally, the positive role of synbiotic supplementation in mental illnesses such as major depressive disorder has been documented. In this case, synbiotics could improve depression symptoms by enhancing tryptophan metabolism and decreasing dopamine metabolite concentrations in the amygdaloid cortex.

It has been suggested that synbiotics could help improve the type and functionality of the microbiota, reduce intestinal inflammation, and promote satiety through increased production of hormones that have this effect on the body. Therefore, this could be beneficial in managing obesity. Synbiotics may play a crucial role in modulating macronutrient metabolism by producing short-chain fatty acids, which bind to G-protein-coupled receptors and increase the secretion of glucagon-like peptide 1 (GLP-1) and peptide YY (PYY) from enteroendocrine L cells. These bindings can trigger insulin production by pancreatic β-cells, inhibit glucagon secretion, decrease hepatic gluconeogenesis, and increase insulin sensitivity. Synbiotics also improve intestinal function, elevate mucin production, and reduce the number of pathogenic gram-negative bacteria in the colon. These changes reduce the transmission of lipopolysaccharides (LPS) across the mucosal wall and metabolic endotoxemia, which may ultimately lead to improvements in insulin receptor function and lower insulin levels. Previous studies have shown that their administration is beneficial for both obesity and typical psychological symptoms of depression or anxiety, among others. A 6-week intervention with synbiotics can significantly reduce depression symptoms compared to a placebo. In this field, a 2017 meta-analysis suggested that probiotics can reduce psychological symptoms, including anxiety, depression, and perceived stress in healthy adult volunteers. The gut microbiota can directly produce neurotransmitters like serotonin and influence its production. It also has immunomodulatory functions and is capable of activating the hypothalamic-pituitary axis through the production of proinflammatory cytokines IL-1 and IL-6.

In this context, an intervention with a synbiotic composed of tannins and beneficial intestinal strains in individuals with obesity could have beneficial effects on health by increasing antioxidant capacity and short-chain fatty acid production, modulating the production of neurotransmitters involved in satiety and mood, and promoting gut microbiota balance, mucosal protection, and improved intestinal permeability.

Therefore, combining synbiotic interventions could provide a synergistic and effective therapy for both metabolic and psychological disorders. Addressing obesity comprehensively, including medical treatment, psychological support for mental health, and synbiotic treatment, could improve emotional state, obesity, and psychological disorders. Ultimately, it could enhance the quality of life for affected individuals. While research in this area is still ongoing and more evidence is needed to understand these interactions underfully, there is growing evidence suggesting that gut microbiota health can influence both physical and mental health in complex and significant ways. Promoting a healthy gut microbiota through a balanced diet, intake of fiber-rich foods and probiotics, as well as stress reduction, may be beneficial for addressing both obesity and psychological disorders, even synergistically with other treatments.

Therefore, our goal is to determine whether the intake of a synbiotic composed of lactic acid bacteria, bifidobacteria, and tannin-based phytocomplexes, is capable of improving anxious and depressive symptoms, glycemic profile, and insulin resistance in patients with obesity, depending on the presence or absence of psychological disorders, through the improvement of the inflammatory profile, appetite control, neurotransmitter production, and the differential alteration of the gut microbiota.

A clinical-basic, prospective, randomized, double-blind, placebo-controlled intervention study is proposed for patients with obesity who present depressive and/or anxiety disorders.

To achieve the proposed objectives, 120 patients with obesity who present depressive and/or anxiety disorders (n=60), and those without disorders (n=60) will be included. The diagnostic criteria for depression and anxiety will be those established in the DSM-5. Furthermore, each group will be randomly divided into 2 subgroups, one of which will receive the synbiotic and the other will receive the corresponding placebo (n=30 per group) for 12 weeks. The randomization process will be carried out using a software program for random assignment. Patients will be enrolled sequentially in the study as they attend the Obesity Unit in the Endocrinology and Nutrition consultations at Dr. Peset Hospital and meet the following criteria:

* Inclusion criteria: patients with a BMI of 30-40 kg/m², aged between 18 and 65 years, with a known disease duration of more than five years. Additionally, all patients will maintain a stable weight (<5% fluctuation) during the 3 months before the study.
* Exclusion criteria: patients who have taken antibiotics 3 months before the start of the study, as well as prior use of supplements containing probiotics and/or prebiotics. Also, patients diagnosed with intestinal diseases, and those who have undergone previous gastrointestinal surgery. Secondary causes of obesity, type 1 diabetes, pregnancy or lactation, active neoplastic disease, and those with established liver or renal failure will be excluded. Finally, patients with other diagnosed psychiatric disorders different from anxiety and/or depression, and those who are undergoing treatment with antidepressants before the start of the study will also be excluded.

Before starting the study, the patients, or their legal representative, will sign an informed consent form after being explained the study's objective and resolving any possible doubts. This study adheres to the ethical guidelines established for human experimentation in Helsinki and its subsequent updates; it will also have approval from the Ethics Committee of the Hospital. The medical information and all data collected during the study will be kept confidential following the Organic Law 15/1999 on Personal Data Protection and the corresponding Royal Decree 1720/07.

At the beginning of the study, the dietitian-nutritionist will carry out an individualized nutritional assessment to calculate the resting energy expenditure and personalized hypocaloric diets will be created, reducing 500 kcal from each individual's total daily energy expenditure, while maintaining the recommended intake of each macronutrient (50-55% carbohydrates, 30-35% fats, and 15% proteins). Dietary monitoring will help avoid bias and reinforce adherence to the diet, along with monitoring side effects. The treatment group will receive a capsule with a synbiotic formulation, and the control group will receive a placebo capsule (maltodextrin), and both groups will be instructed to take it daily for 12 weeks. The synbiotic will consist of a probiotic part composed of Lactobacillus acidophilus, Lactobacillus casei, and Bifidobacterium lactis (2×10⁹ CFU/g each), and a prebiotic part composed of phytocomplexes based on tannins (350 mg) extracted from various sources. The placebo will look identical to the synbiotic capsule. To maintain blinding for the staff participating in the trial, the preparation of the study products and the filling of the containers will be done by the companies SILVATEAM and SACCO, which will operate under unblinded conditions.

At the beginning of the intervention, a structured psychological interview will be conducted to gather information about the patient's current condition; history and evolution of the disease (obesity and psychological disorder), eating patterns, sleep quality, associated psychological comorbidities, family and social areas, motivation for change, and expectations. The impact of obesity on the patient's quality of life (emotional, social, and personal) will be evaluated. Psychological follow-up will take place at 4, 6, and 12 weeks of the study. During the interventions, motivation status, eating habits, lifestyle, self-control, cognitive-behavioral change, and relapse prevention will be assessed.

At the beginning of the study and after the dietary intervention, fasting blood samples (12 hours), saliva, urine (24 hours), and stool samples will be collected. The following parameters will be determined:

1. Anthropometric Parameters and Body Composition Weight and height will be measured, and BMI will be calculated (weight / (height)²). Waist and hip circumference, as well as blood pressure, will also be determined. Additionally, a vector analysis using bioelectrical impedance (seca mBCA 550®) will be performed both at the beginning and the end of the intervention.

   Patients will complete a 3-day dietary log (including 1 weekend day) at the beginning, 6 weeks, and 12 weeks, along with the IPAQ questionnaire to monitor physical activity. They will also complete a questionnaire on product adherence and compliance, and if they have experienced any adverse effects after taking the product.
2. Psychological Evaluation First, the investigators will apply the Depression Anxiety and Stress Scale 21 (DASS-21) questionnaire. Based on the initial results, stress, anxiety, and depression will be evaluated using three validated scales: the Beck Depression Inventory (BDI-2), the Perceived Stress Scale (PSS), the State-Trait Anxiety Inventory (STAI), and self-esteem using the Rosenberg questionnaire. This evaluation will allow the subject's classification into both groups (obesity with and without anxiety and/or depression), and check if there is a significant improvement after the synbiotic intake group.
3. Biochemical Parameters A complete lipid profile will be assessed, determining total cholesterol (TC) and triglycerides (TG) using enzymatic methods, HDL-C (direct precipitation method), LDL-C (calculated using Friedewald's formula), and VLDL-C (TG/5). Apolipoproteins B and A-I will be determined by nephelometry. Non-HDL cholesterol (TC-HDL) and the atherogenic plasma index (API = log (TG/HDL)) will be calculated. Fasting blood glucose and insulin will be measured using the hexokinase enzymatic method and chemiluminescence, respectively, and the HOMA index will be calculated to assess insulin resistance. Liver and kidney function, complete blood count, coagulation, and hormonal profile will be evaluated using the following markers: AST, ALT, GGT, LDH, alkaline phosphatase, creatinine, glomerular filtration rate, A1c, and thyroid function (TSH, free T4). All of these parameters will be determined in the Clinical Analysis Service of the Dr. Peset University Hospital.
4. Biomarker Determination d.1) Inflammatory Parameters and Antioxidant Capacity The inflammatory state will be assessed by determining the concentrations of ultrasensitive C-reactive protein, IL6, TNF, IL1b, adiponectin, PAI-1, and IL10, using Luminex xMAP-Multiplex technology. Sample processing and data analysis will be performed following the manufacturer's instructions. Serum levels of LPS will be determined by ELISA. Total antioxidant capacity in serum will be determined using the E-BQC system (Bioquochem).

d.2) Determination of Peptides and Intestinal Function Serum levels of intestinal hormones (GIP, GLP1, PYY, ghrelin, leptin, CCK) will be determined using Luminex X-MAP technology. To evaluate intestinal permeability and microbial translocation, plasma levels of zonulin, occludin, LBP, FABP2/I-FABP, and Reg3A will be measured using ELISA Kits. Detection of β-glucan in plasma will be performed using the Limulus Amebocyte Lysate (LAL) assay.

d.3) Neurotransmitter Peptide Analysis Cortisol, dopamine, serotonin, and oxytocin levels in plasma, 24-hour urine, or saliva will be determined using ELISA kits or Luminex X-MAP technology.

d.4) Metabolomic Analysis NMR (Nuclear Magnetic Resonance) will be applied to obtain extensive metabolic profiles from large, well-phenotyped patient cohorts. Initially, all samples will be analyzed by NMR, obtaining a global metabolic profile of up to 40 metabolites including amino acids, sugars, phospholipids, inflammation markers, glycoproteins, lipoparticles, and some microbial co-metabolites.

The statistical significance of the different metabolites will be analyzed using covariance tests corrected for potential false discovery rate (FDR) using SPSS and Matlab software. Chemometric analysis to construct diagnostic, classification and predictive models will be performed using custom Matlab scripts and PLS Toolbox for PCA, projection to latent structure-discriminant analysis (PLS-DA), hierarchical cluster analysis (HCA), and similar approaches on spectral data to classify groups based on clinical and intervention parameters. Metabolic networks will be built using CytoScape and the Kyoto Encyclopedia of Genes and Genomes (KEGG) for genomics, integrating metabolomic results and other molecular outcomes of the project. Finally, all results will be evaluated through cross-validation, and the discriminatory/predictive power of the different metabolites and scores will be analyzed using receiver operating characteristic (ROC) curves.

d.5) Study of the Microbiota Nucleic acid purification, 16S rRNA gene amplification, and sequencing First, the stool samples will be triturated, homogenized, and lysed using a Fastprep system (MP Biomedicals). Total DNA will be extracted following the automated Magna Pure LC protocol (Roche, Manheim, Germany) according to the manufacturer's instructions. Metagenomic libraries will be obtained using the NEXTERA XT kit following Illumina's protocol. The V3-V4 regions of the 16S rRNA will be amplified, and the libraries will be purified following Illumina's protocol.

MiSeq sequencing will be performed using the V3 kit (2x300 cycles), generating 300-bp reads every 65 hours, starting from each end of the amplicon. Ultra-deep sequencing will be performed using an Illumina sequencer at the FISABIO-Salud Pública Center.

Phylogenetic analysis of 16S rRNA will be carried out using QIIME software. Functional assignment of metagenomic reads will be performed using dedicated bioinformatics pipelines developed at FISABIO (integrating cutting-edge methodologies in the field with customizable scripts).

Microbial community analyses (biodiversity, clustering, heat maps) and statistical analysis will be performed using R software. For biomarker discovery analysis, the LEfSe platform will be used.

d.6) Gene Expression Analysis Changes in gene expression levels will be evaluated using Nanostring® technology for nCounter®, which will allow us to identify messenger molecules that are altered between obese patients with/without psychological disorders. This system enables the hybridization of each target molecule with a fluorescent probe for individual identification without retrotranscription or amplification, using minimal sample amounts. Total RNA will be extracted from PBMCs using the GeneAll® RibospinTM total kit, and from just 100-200 ng of total RNA, the multiplex metabolism panel will assess 768 genes, focusing on inflammatory and metabolic pathways. The results will be analyzed using the nSolver tool. These experiments will be subcontracted to Diagnostica Longwood, S.L.

d.7) In Vitro Study of the Mechanism of Action of Colonic Digestate on Complex Cellular Models Simulating the Gut-Brain Axis The use and design of an organ-on-chip (OoC) model is proposed, with intestinal cells in contact with the fermentation digestate (from patient feces) and neuroblastoma cells in contact with the absorbed material, specifically designed to study the mechanism of action of the synbiotic. For biomarker analysis, changes at the intestinal level in inflammatory cytokines and neuronal cell receptor changes will be observed, which can later be related to the in vivo results. The design will include obtaining sufficient control sample replicates, with colonic digestate after stabilization, and with colonic digestate after treatment with placebo or synbiotic.

ELIGIBILITY:
Inclusion Criteria:

* Patients with BMI 30-40kg/m2, with at least 5 years of diagnosed obesity evolution.
* Patients have had stable body weight (<5% of body weight changes) during the 3 months prior to the study.
* Participants between 18 and 65 years of age.

Exclusion Criteria:

* All patients with acute or chronic inflammatory diseases, neoplasic disease, secondary causes of obesity (uncontrolled hypothyroidism, Cushing's syndrome), or established liver and kidney failure (according to transaminase levels ±2 SD of the mean and estimated glomerular filtration rate using the CKD-EPI formula >60), previous bariatric surgery, and women during pregancy or lactation, will be excluded.
* Participants who have been treated with antibiotics 3 months prior to inclusion.
* Patients with different psychiatric disorders apart from anxiety and/or depression, and also those who are already on antidepressants before the inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Analyze the changes in the diversity of the intestinal microbiota after the symbiotic intake. | 3 years
  To assess the alpha-diversity of the intestinal microbiota after the symbiotic intake, defined as the average diversity of species in an ecosystem, the Shannon index will be used. The results are interpreted as follows: values less than 2 are considered low in diversity and values greater than 3 are high in species diversity.
Evaluate the differences in the diversity of the intestinal microbiota depending on whether participants have received the synbiotic or the placebo supplement. | 3 years
  To assess the alpha-diversity of the intestinal microbiota, defined as the average diversity of species in an ecosystem, the Shannon index will be used. A significant difference between both groups (synbiotic and placebo) will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Identify and assess the differences in metabolic pathways of gut microbiota after the synbiotic intake. | 3 years
  Genetic markers of inflammation and metabolic pathways will be analyzed from the faeces samples, in order to identify different clusters of these pathways and determine the potential functions of gut microbiota. For that purpose, transcriptome will be quantified with nanostring techology. The relative quantity of gene expression (fold change) of each gene will be calculated with the comparative 2-ΔΔCT method, and significant differences will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval.
Assess if there is a significant improvement in psychological parameters of anxiety and depression after the synbiotic intake. | 3 years
  Psychological parameters will include anxiety and depression symptoms. Anxiety and depression will be quantified using a validated scale called Depression Anxiety and Stress Scale 21 (DASS-21), which focuse on psychological symptoms and to diagnose both anxiety and depression disorders. In this scale, in depression questions, a score of 0-9 indicates normality, 10-13 mild depression, 14-20 moderate depression, 21-27 severe depression, and >27 extreme severe depression; in anxiety scale, a score of 0-7 reflects normality, 8-9 mild anxiety, 10-14 moderate, 15-19 severe, and >19 extreme severe anxiety; in stress scale, a score of 0-14 indicates normality, 15-18 mild stress, 19-25 moderate stress, 26-33 severe stress, and >33 extreme severe stress.

SECONDARY OUTCOMES:
Evaluate significant changes in body fat mass percentage after the synbiotic intake. | 3 years
  Percentage of body fat mass will be measured by bioelectrical impedance. It is considered to be high when ≥25% in men and ≥30% in women. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval. Synbiotic group will be compared to placebo group to check if there are also significant differences (p-value <0.05 with a 95% confidence interval between both mean values).
Assess significant changes in high-sensitivity C-reactive protein (hs-CRP) as an inflammatory parameter after the synbiotic intake | 3 years
  Participants will be considered to have achieved an improvement in high-sensitivity C-reactive protein levels if they normalize its value (normality values defined between 0 and 1.69mg/dl). Synbiotic group will be compared to placebo group to check if there are also significant differences (p-value <0.05 with a 95% confidence interval between both mean values).
Evaluate significant changes in C3 protein as an inflammatory parameter after the synbiotic intake. | 3 years
  Participants will be considered to have achieved an improvement in C3 protein if they normalize its value (normality values defined between 81 and 157mg/dl). Results in synbiotic group will be compared to placebo group to check if there are significant differences between both groups (p-value <0.05 with a 95% confidence interval between both mean values).
Assess significant changes in plasmatic homocysteine as an inflammatory parameter after the synbiotic intake. | 3 years
  Participants will be considered to have achieved an improvement in plasmatic homocysteine if they normalize its value (normality values defined between 5 and 15µmol/L). Synbiotic group will be compared to placebo group to check if there are also significant differences (p-value <0.05 with a 95% confidence interval between both mean values).
Evaluate significant changes in interleukin 1-beta (IL-1B) levels as a pro-inflammatory molecule after the synbiotic intake | 3 years
  IL-1B levels will be measured using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval. Significant differences between both groups (synbiotic and placebo) will be assessed (p-value <0.05 with a 95% confidence interval between both mean values).
Evaluate significant changes in interleukin 6 (IL-6) levels as a pro-inflammatory molecule after the synbiotic intake. | 3 years
  IL-6 levels will be measured using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval. Results in synbiotic group will be compared to placebo group to check if there are significant differences between both groups (p-value <0.05 with a 95% confidence interval between both mean values).
Evaluate significant changes in tumor necrosis factor alpha (TNF-alpha) levels as a pro-inflammatory molecule after the synbiotic intake. | 3 years
  TNF-alpha levels will be measured using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval. Results in synbiotic group will be compared to placebo group to check if there are significant differences between both groups (p-value <0.05 with a 95% confidence interval between both mean values).
Assess significant changes in superoxide dismutase (SOD) levels after the synbiotic intake. | 3 years
  Superoxide dismutase levels will be measured using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval. Results will be compared between both groups (synbiotic and placebo) to evaluate if there are significant differences (p-value <0.05 with a 95% confidence interval between both mean values).
Evaluate if there is a significant reduction after the synbiotic intake in total ROS levels. | 3 years
  Total ROS levels will be assessed by a flow cytometry assay. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval. Significant differences between both groups (synbiotic and placebo) will be assessed (p-value <0.05 with a 95% confidence interval between both mean values).
Assess if there is a significant reduction after the synbiotic intake in glutathione levels. | 3 years
  Total glutathione levels will be assessed by a flow cytometry assay. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval. Results in synbiotic group will be compared to placebo group to check if there are significant differences between both groups (p-value <0.05 with a 95% confidence interval between both mean values).
Analyze if there is a significant change after the synbiotic intake in total free radicals and superoxide levels. | 3 years
  Total free radicals and superoxide content will be assessed by a flow cytometry assay. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval. Results in synbiotic group will be compared to placebo group to check if there are significant differences between both groups (p-value <0.05 with a 95% confidence interval between both mean values).
Analyze if there is a significant reduction after the synbiotic intake in mitochondrial ROS production. | 3 years
  Mitochondrial ROS production will be assessed by a flow cytometry assay. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval. Results will be compared between both groups (synbiotic and placebo) to evaluate if there are significant differences (p-value <0.05 with a 95% confidence interval between both mean values).
Analyze the significant differences between metabolomic profile in faeces before and after the synbiotic supplementation.. | 3 years
  NMR spectra will be used to obtain spectra from serum samples from the cohort. In order to evaluate if there will be significant differences after the dietetic intervention, a PLS-DA model for discrimination between basal and post intervention levels will be performed. Scores plots will be calculated with a 95% confidence interval. Synbiotic group will be compared to placebo group to check if there are also significant differences (p-value <0.05 with a 95% confidence interval between both mean values).
Analyze if there is a significant reduction after the synbiotic intake in adipsin levels. | 3 years
  Adipsin levels will be measured using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval. Synbiotic group will be compared to placebo group to check if there are also significant differences (p-value <0.05 with a 95% confidence interval between both mean values).
Assess significant changes in plasmatic resistin levels as an inflammatory parameter after the synbiotic intervention. | 3 years
  Resistin levels will be measured using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval. Synbiotic group will be compared to placebo group to check if there are also significant differences (p-value <0.05 with a 95% confidence interval between both mean values).
Evaluate significant reductions in Plasminogen activator inhibitor-1 (PAI-1) as an inflammatory parameter after the synbiotic intake. | 3 years
  PAI-1 levels will be measured using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval. Synbiotic group will be compared to placebo group to check if there are also significant differences (p-value <0.05 with a 95% confidence interval between both mean values).
Evaluate if there is a significant reduction after the synbiotic intake in Lipopolysaccharide (LPS) serum levels. | 3 years
  LPS levels will be measured using ELISA kits. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval. Synbiotic group will be compared to placebo group to check if there are also significant differences (p-value <0.05 with a 95% confidence interval between both mean values).
Evaluate significant changes in lipopolysaccharide-binding protein (LBP) levels as a pro-inflammatory biomarker after the synbiotic intake. | 3 years
  LBP levels will be measured using ELISA kits. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval. Synbiotic group will be compared to placebo group to check if there are also significant differences (p-value <0.05 with a 95% confidence interval between both mean values).
Evaluate if there is a significant change in Regenerating islet-derived protein 3 alpha (REG3A) levels after the synbiotic supplementation. | 3 years
  REG3A levels will be assessed by ELISA kits. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval. Synbiotic group will be compared to placebo group to check if there are also significant differences (p-value <0.05 with a 95% confidence interval between both mean values).
Assess if there is a significant reduction after the synbiotic intake in zonulin levels. | 3 years
  Zonulin levels will be assessed by ELISA kits. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval. Synbiotic group will be compared to placebo group to check if there are also significant differences (p-value <0.05 with a 95% confidence interval between both mean values).
Analyze if there is a significant change after the synbiotic intake in leptin and ghrelin levels. | 3 years
  Both leptin and ghrelin levels will be assessed using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval. Synbiotic group will be compared to placebo group to check if there are also significant differences (p-value <0.05 with a 95% confidence interval between both mean values).
Assess significant changes in serum Glucagon-like peptide-1 (GLP-1) and Gastric inhibitory polypeptide (GIP) levels after the synbiotic intake. | 3 years
  GLP-1 and GIP levels will be assessed using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval. Synbiotic group will be compared to placebo group to check if there are also significant differences (p-value <0.05 with a 95% confidence interval between both mean values).
Assess if there is a significant improvement after the synbiotic intake in peptide YY (PYY) and cholecystokinin (CCK) levels. | 3 years
  PYY and CCK levels will be assessed using the Luminex® 200 analyzer system. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval. Synbiotic group will be compared to placebo group to check if there are also significant differences (p-value <0.05 with a 95% confidence interval between both mean values).
Evaluate if there is a significant improvement in ocludin and Fatty acid-binding protein 2 (FABP2 or I-FABP) levels, as biomarkers of gut permeability. | 3 years
  Ocludin and FABP2 levels will be assessed using ELISA kits. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval. Synbiotic group will be compared to placebo group to check if there are also significant differences (p-value <0.05 with a 95% confidence interval between both mean values).
Assess if there is a significant reduction after the symbiotic intake in neurotransmitter levels. | 3 years
  Levels of cortisol, dopamine, serotonin and oxytocin in plasma, 24-hour urine or saliva will be measured using ELISA kits or X-MAP technology Luminex. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval. Synbiotic group will be compared to placebo group to check if there are also significant differences (p-value <0.05 with a 95% confidence interval between both mean values).
Analyze if there is a significant reduction after the symbiotic intake in β-D-Glucan (BDG) levels as a biomarker of impaired gut permeability. | 3 years
  BDG levels will be assessed by the Limulus amebocyte lysate (LAL) assay. A significant improvement will be considered when notable differences are observed in the mean values between groups measured through p-value (<0.05) with a 95% confidence interval. Synbiotic group will be compared to placebo group to check if there are also significant differences (p-value <0.05 with a 95% confidence interval between both mean values).

CONTACTS AND LOCATIONS:
Locations (1):
- FISABIO, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hou K, Wu ZX, Chen XY, Wang JQ, Zhang D, Xiao C, Zhu D, Koya JB, Wei L, Li J, Chen ZS. Microbiota in health and diseases. Signal Transduct Target Ther. 2022 Apr 23;7(1):135. doi: 10.1038/s41392-022-00974-4. PMID 35461318
- [Background] Molino S, Pilar Francino M, Angel Rufian Henares J. Why is it important to understand the nature and chemistry of tannins to exploit their potential as nutraceuticals? Food Res Int. 2023 Nov;173(Pt 2):113329. doi: 10.1016/j.foodres.2023.113329. Epub 2023 Jul 27. PMID 37803691
- [Background] Rusch JA, Layden BT, Dugas LR. Signalling cognition: the gut microbiota and hypothalamic-pituitary-adrenal axis. Front Endocrinol (Lausanne). 2023 Jun 19;14:1130689. doi: 10.3389/fendo.2023.1130689. eCollection 2023. PMID 37404311
- [Background] Sanlier N, Kocabas S. The effect of probiotic, prebiotic and gut microbiota on ASD: A review and future perspectives. Crit Rev Food Sci Nutr. 2023;63(15):2319-2330. doi: 10.1080/10408398.2021.1973957. Epub 2021 Sep 6. PMID 34486891
- [Background] Oraphruek P, Chusak C, Ngamukote S, Sawaswong V, Chanchaem P, Payungporn S, Suantawee T, Adisakwattana S. Effect of a Multispecies Synbiotic Supplementation on Body Composition, Antioxidant Status, and Gut Microbiomes in Overweight and Obese Subjects: A Randomized, Double-Blind, Placebo-Controlled Study. Nutrients. 2023 Apr 13;15(8):1863. doi: 10.3390/nu15081863. PMID 37111082
- [Background] Ng QX, Lim YL, Yaow CYL, Ng WK, Thumboo J, Liew TM. Effect of Probiotic Supplementation on Gut Microbiota in Patients with Major Depressive Disorders: A Systematic Review. Nutrients. 2023 Mar 10;15(6):1351. doi: 10.3390/nu15061351. PMID 36986088
- [Background] Tamtaji OR, Taghizadeh M, Daneshvar Kakhaki R, Kouchaki E, Bahmani F, Borzabadi S, Oryan S, Mafi A, Asemi Z. Clinical and metabolic response to probiotic administration in people with Parkinson's disease: A randomized, double-blind, placebo-controlled trial. Clin Nutr. 2019 Jun;38(3):1031-1035. doi: 10.1016/j.clnu.2018.05.018. Epub 2018 Jun 1. PMID 29891223
- [Background] Fox M, Knorr DA, Haptonstall KM. Alzheimer's disease and symbiotic microbiota: an evolutionary medicine perspective. Ann N Y Acad Sci. 2019 Aug;1449(1):3-24. doi: 10.1111/nyas.14129. Epub 2019 Jun 10. PMID 31180143
- [Background] Fernandes R, do Rosario VA, Mocellin MC, Kuntz MGF, Trindade EBSM. Effects of inulin-type fructans, galacto-oligosaccharides and related synbiotics on inflammatory markers in adult patients with overweight or obesity: A systematic review. Clin Nutr. 2017 Oct;36(5):1197-1206. doi: 10.1016/j.clnu.2016.10.003. Epub 2016 Oct 8. PMID 27771020
- [Background] Rabiei S, Hedayati M, Rashidkhani B, Saadat N, Shakerhossini R. The Effects of Synbiotic Supplementation on Body Mass Index, Metabolic and Inflammatory Biomarkers, and Appetite in Patients with Metabolic Syndrome: A Triple-Blind Randomized Controlled Trial. J Diet Suppl. 2019;16(3):294-306. doi: 10.1080/19390211.2018.1455788. Epub 2018 Apr 19. PMID 29672196
- [Background] Hadi A, Mohammadi H, Miraghajani M, Ghaedi E. Efficacy of synbiotic supplementation in patients with nonalcoholic fatty liver disease: A systematic review and meta-analysis of clinical trials: Synbiotic supplementation and NAFLD. Crit Rev Food Sci Nutr. 2019;59(15):2494-2505. doi: 10.1080/10408398.2018.1458021. Epub 2018 Apr 20. PMID 29584449
- [Background] Hadi A, Alizadeh K, Hajianfar H, Mohammadi H, Miraghajani M. Efficacy of synbiotic supplementation in obesity treatment: A systematic review and meta-analysis of clinical trials. Crit Rev Food Sci Nutr. 2020;60(4):584-596. doi: 10.1080/10408398.2018.1545218. Epub 2018 Dec 30. PMID 30595036
- [Background] Mohammadi H, Ghavami A, Hadi A, Askari G, Symonds M, Miraghajani M. Effects of pro-/synbiotic supplementation on anthropometric and metabolic indices in overweight or obese children and adolescents: A systematic review and meta-analysis. Complement Ther Med. 2019 Jun;44:269-276. doi: 10.1016/j.ctim.2019.05.008. Epub 2019 May 8. PMID 31126565
- [Background] Zhao Z, Xiao G, Xia J, Guo H, Yang X, Jiang Q, Wang H, Hu J, Zhang C. Effectiveness of probiotic/prebiotic/synbiotic treatments on anxiety: A systematic review and meta-analysis of randomized controlled trials. J Affect Disord. 2023 Dec 15;343:9-21. doi: 10.1016/j.jad.2023.09.018. Epub 2023 Sep 20. PMID 37734624
- [Background] Taverniti V, Koirala R, Dalla Via A, Gargari G, Leonardis E, Arioli S, Guglielmetti S. Effect of Cell Concentration on the Persistence in the Human Intestine of Four Probiotic Strains Administered through a Multispecies Formulation. Nutrients. 2019 Jan 29;11(2):285. doi: 10.3390/nu11020285. PMID 30699901
- [Background] Ozdal T, Sela DA, Xiao J, Boyacioglu D, Chen F, Capanoglu E. The Reciprocal Interactions between Polyphenols and Gut Microbiota and Effects on Bioaccessibility. Nutrients. 2016 Feb 6;8(2):78. doi: 10.3390/nu8020078. PMID 26861391
- [Background] Marrone G, Di Lauro M, Izzo F, Cornali K, Masci C, Vita C, Occhiuto F, Di Daniele N, De Lorenzo A, Noce A. Possible Beneficial Effects of Hydrolyzable Tannins Deriving from Castanea sativa L. in Internal Medicine. Nutrients. 2023 Dec 22;16(1):45. doi: 10.3390/nu16010045. PMID 38201875
- [Background] Li Y, Zhu L, Guo C, Xue M, Xia F, Wang Y, Jia D, Li L, Gao Y, Shi Y, He Y, Yuan C. Dietary Intake of Hydrolyzable Tannins and Condensed Tannins to Regulate Lipid Metabolism. Mini Rev Med Chem. 2022;22(13):1789-1802. doi: 10.2174/1389557522666211229112223. PMID 34967286
- [Background] Molino S, Casanova NA, Rufian Henares JA, Fernandez Miyakawa ME. Natural Tannin Wood Extracts as a Potential Food Ingredient in the Food Industry. J Agric Food Chem. 2020 Mar 11;68(10):2836-2848. doi: 10.1021/acs.jafc.9b00590. Epub 2019 Jun 3. PMID 31117489
- [Background] Zhang Q, Chen B, Zhang J, Dong J, Ma J, Zhang Y, Jin K, Lu J. Effect of prebiotics, probiotics, synbiotics on depression: results from a meta-analysis. BMC Psychiatry. 2023 Jun 29;23(1):477. doi: 10.1186/s12888-023-04963-x. PMID 37386630
- [Background] Xiao H, Kang S. The Role of the Gut Microbiome in Energy Balance With a Focus on the Gut-Adipose Tissue Axis. Front Genet. 2020 Apr 7;11:297. doi: 10.3389/fgene.2020.00297. eCollection 2020. PMID 32318095
- [Background] Liu BN, Liu XT, Liang ZH, Wang JH. Gut microbiota in obesity. World J Gastroenterol. 2021 Jul 7;27(25):3837-3850. doi: 10.3748/wjg.v27.i25.3837. PMID 34321848
- [Background] Wadden TA, Tronieri JS, Butryn ML. Lifestyle modification approaches for the treatment of obesity in adults. Am Psychol. 2020 Feb-Mar;75(2):235-251. doi: 10.1037/amp0000517. PMID 32052997
- [Background] Chen M, Ruan G, Chen L, Ying S, Li G, Xu F, Xiao Z, Tian Y, Lv L, Ping Y, Cheng Y, Wei Y. Neurotransmitter and Intestinal Interactions: Focus on the Microbiota-Gut-Brain Axis in Irritable Bowel Syndrome. Front Endocrinol (Lausanne). 2022 Feb 16;13:817100. doi: 10.3389/fendo.2022.817100. eCollection 2022. PMID 35250873
- [Background] Asadi A, Shadab Mehr N, Mohamadi MH, Shokri F, Heidary M, Sadeghifard N, Khoshnood S. Obesity and gut-microbiota-brain axis: A narrative review. J Clin Lab Anal. 2022 May;36(5):e24420. doi: 10.1002/jcla.24420. Epub 2022 Apr 14. PMID 35421277
- [Background] Boulange CL, Neves AL, Chilloux J, Nicholson JK, Dumas ME. Impact of the gut microbiota on inflammation, obesity, and metabolic disease. Genome Med. 2016 Apr 20;8(1):42. doi: 10.1186/s13073-016-0303-2. PMID 27098727
- [Background] Strawbridge R, Young AH, Cleare AJ. Biomarkers for depression: recent insights, current challenges and future prospects. Neuropsychiatr Dis Treat. 2017 May 10;13:1245-1262. doi: 10.2147/NDT.S114542. eCollection 2017. PMID 28546750
- [Background] Du Y, Gao XR, Peng L, Ge JF. Crosstalk between the microbiota-gut-brain axis and depression. Heliyon. 2020 Jun 3;6(6):e04097. doi: 10.1016/j.heliyon.2020.e04097. eCollection 2020 Jun. PMID 32529075
- [Background] Rutsch A, Kantsjo JB, Ronchi F. The Gut-Brain Axis: How Microbiota and Host Inflammasome Influence Brain Physiology and Pathology. Front Immunol. 2020 Dec 10;11:604179. doi: 10.3389/fimmu.2020.604179. eCollection 2020. PMID 33362788
- [Background] Alli SR, Gorbovskaya I, Liu JCW, Kolla NJ, Brown L, Muller DJ. The Gut Microbiome in Depression and Potential Benefit of Prebiotics, Probiotics and Synbiotics: A Systematic Review of Clinical Trials and Observational Studies. Int J Mol Sci. 2022 Apr 19;23(9):4494. doi: 10.3390/ijms23094494. PMID 35562885
- [Background] McKean J, Naug H, Nikbakht E, Amiet B, Colson N. Probiotics and Subclinical Psychological Symptoms in Healthy Participants: A Systematic Review and Meta-Analysis. J Altern Complement Med. 2017 Apr;23(4):249-258. doi: 10.1089/acm.2016.0023. Epub 2016 Nov 14. PMID 27841940
- [Background] Sarwer DB, Polonsky HM. The Psychosocial Burden of Obesity. Endocrinol Metab Clin North Am. 2016 Sep;45(3):677-88. doi: 10.1016/j.ecl.2016.04.016. PMID 27519139
- [Background] Steptoe A, Frank P. Obesity and psychological distress. Philos Trans R Soc Lond B Biol Sci. 2023 Oct 23;378(1888):20220225. doi: 10.1098/rstb.2022.0225. Epub 2023 Sep 4. PMID 37661745
- [Background] Namazi N, Atlasi R, Aletaha A, Asadi M, Larijani B. Trend of nutrition research in endocrine disorders, gaps, and future plans: a collection of experiences of an endocrinology research institute. J Diabetes Metab Disord. 2021 Jan 22:1-8. doi: 10.1007/s40200-020-00707-w. Online ahead of print. PMID 33500881
- [Background] Bluher M, Aras M, Aronne LJ, Batterham RL, Giorgino F, Ji L, Pietilainen KH, Schnell O, Tonchevska E, Wilding JPH. New insights into the treatment of obesity. Diabetes Obes Metab. 2023 Aug;25(8):2058-2072. doi: 10.1111/dom.15077. Epub 2023 May 5. PMID 37055715
- [Background] Lin X, Li H. Obesity: Epidemiology, Pathophysiology, and Therapeutics. Front Endocrinol (Lausanne). 2021 Sep 6;12:706978. doi: 10.3389/fendo.2021.706978. eCollection 2021. PMID 34552557